CLINICAL TRIAL: NCT05692817
Title: Evaluation of Maxillary Canine Retraction Assisted With Two Different Methods of Low-Intensity Pulsed Ultrasound: A Controlled Clinical Study
Brief Title: Evaluation of Maxillary Canine Retraction Assisted With Two Different Methods of Low-Intensity Pulsed Ultrasound
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ammar Kasem Alzoubi (Other)
Responsible Party: Sponsor-Investigator, Ammar Kasem Alzoubi, Dentist, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 891/2786
Record Dates: First submitted 2023-01-12; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Orthodontic Appliance Complication

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- one- weeks group (Experimental)
  Interventions: Device: Low-Intensity Pulsed Ultrasound
- three-weeks group (Experimental)
  Interventions: Device: Low-Intensity Pulsed Ultrasound

INTERVENTIONS:
Device: Low-Intensity Pulsed Ultrasound — The total sample will be randomly divided into two equal groups (according to method of application of the lipus on the intervention side)as follows: ■ Group I: will include 8 patients who will receive lipus with maxillary canine retraction that will be performed every (3 weeks) on intervention 6 sides according to a standardized protocol.
  ▪ Group II: will include 8 patients who will receive lipus that will be performed every (1 week) on intervention sides according to a standardized protocol.

SUMMARY:
The current clinical study will be done for evaluation of maxillary canine retraction assisted with application of two different methods of low-intensity pulsed ultrasound.

ELIGIBILITY:
Inclusion Criteria:

-

All patients should satisfy the following criteria:

1. An age ranges from 15-22 years.
2. Severe crowding or protrusion requiring 1st premolar extractions followed by symmetrical canine retraction.
3. All permanent teeth present, 3rd molars are excluded.
4. Good oral hygiene.
5. No systemic disease/medication that could interfere with orthodontic tooth Movement (OTM).
6. No previous orthodontic treatment.

Exclusion Criteria:

* 1. Patient diagnosed to have an indication for non-extraction approach. 2. Poor oral hygiene or periodontally compromised patient. 5 3. Patient with craniofacial anomalies or previous history of trauma, bruxism or parafunctions. 4. Previous orthodontic treatment. 5. Any implanted assistive devices (e.g., pacemakers, cochlear implants, etc.) 6. Pregnant females.

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of canine retraction | four months
  distance

CONTACTS AND LOCATIONS:
Locations (1):
- Alazhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided